CLINICAL TRIAL: NCT00460720
Title: Compliance Survey of ADHD Medication for Optimal Satisfaction (COSMOS)
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Medical Director, Johnson & Johnson Taiwan Ltd
Other Study IDs: CR013384
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Methylphenidate; MPH; Extended-Release Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Observational treatment compliance survey

INTERVENTIONS:
Other: Observational treatment compliance survey — Observational treatment compliance survey

SUMMARY:
The survey is designed to identify non-compliant Attention Deficit Hyperactivity Disorder (ADHD) patients who are currently on Immediate- Released Methylphenidate (IR-MPH) and observe any change in compliance after treating with other drugs intended to treat ADHD for over 3 weeks

DETAILED DESCRIPTION:
This is an Observational, survey study. The survey is designed to be administered in two stages. In the first stage, patients who were prescribed Immediate-Released Methylphenidate (IR-MPH) for over 3 months, who are also on IR-MPH 1 month prior and who meet inclusion criteria will be enrolled. On survey day 1, the patients, parents/caregivers, and clinicians will assess patient drug compliance. For patients considered non-compliant, the Investigator will decide whether or not to change current medication. Those patients whose medication is changed from IR-MPH to another treatment for ADHD, will be enrolled into the second stage. On survey day 1, Clinical Global Impression (CGI) and the effects of the medication on sleep quality, decreased appetite, dizziness and or headache, and gastrointestinal upset will be assessed based on clinical interview. Any other side effects shown during medication treatment will be also recorded in the first stage. Parent/Caregivers will need to complete the Swanson, Nolan and Pelham (SNAP) Questionnaire which will evaluate the ADHD child's symptoms of inattention, hyperactivity, impulsivity and oppositional defiant disorder. In the second stage, those ADHD patients who meet the definition of non-compliance will be treated with other medications for over three weeks. On the first visit back after starting treatment with other medications, drug compliance, CGI, any change in negative parent-child interaction, overall classroom behavior, overall academic performance, the effects on sleep quality, decreased appetite, diziness and or headache, and gastrointestinal upset will be assessed by Investigator interview. Parent/Caregivers will need to complete SNAP Questionaire which will evaluate the ADHD child's symptoms of inattention, hyperactivity, impulsivity and oppositional defiant disorder. It is a survey type of study. No study drug has been used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of DSM-IV ADHD
* Patients were previously treated with Immediate-Released Methylphenidate (IR-MPH) taken once a day, twice a day, three times a day, or four times a day over three months and who were also on IR-MPH the last month without severe adverse events or possible contraindications with MPH
* Patients whose parent or guardian has signed and dated an informed consent to participate in the survey of drug compliance
* Patients who are still at school

Exclusion Criteria:

* ADHD patients who have systematic disease or clinically significant gastrointestinal problems, including narrowing (pathologic or iatrogenic) of the gastrointestinal tract
* ADHD patients also diagnosed with psychosis except for Conduct Disorder and Oppositional Defiant Disorder

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 6-16 years old with clinical diagnosis of DSM-IV ADHD
Sampling Method: Probability Sample
Enrollment: 591 (Actual)
Dates: Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The change from survey day 1 to first visit in Clinical Global Impression score | 3 weeks

SECONDARY OUTCOMES:
The change from baseline in Swanson, Nolan and Pelham (SNAP) Questionnaire. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

REFERENCES:
- [Derived] Chou WJ, Chou MC, Tzang RF, Hsu YC, Gau SS, Chen SJ, Wu YY, Huang YF, Liang HY, Cheng H. Better efficacy for the osmotic release oral system methylphenidate among poor adherents to immediate-release methylphenidate in the three ADHD subtypes. Psychiatry Clin Neurosci. 2009 Apr;63(2):167-75. doi: 10.1111/j.1440-1819.2009.01937.x. PMID 19335386
- [Derived] Gau SS, Chen SJ, Chou WJ, Cheng H, Tang CS, Chang HL, Tzang RF, Wu YY, Huang YF, Chou MC, Liang HY, Hsu YC, Lu HH, Huang YS. National survey of adherence, efficacy, and side effects of methylphenidate in children with attention-deficit/hyperactivity disorder in Taiwan. J Clin Psychiatry. 2008 Jan;69(1):131-40. doi: 10.4088/jcp.v69n0118. PMID 18312048